Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)



"To Save A Life Is To Save A Universe"

Protocol Identifying Number: AML003 Study Name: ARMADA 2000

**IND Number: 114-372** 

**EudraCT Number: 2018-001588-22** 

**IND Sponsor: Rafael Pharmaceuticals Inc.** 

1 Duncan Drive Cranbury, NJ 08512-3629

Version Number: 8.00 Amendment 5.0

October 19th, 2020

Superseded Version:
Version 7.0, August 17<sup>th</sup>, 2020
Version 6.0, April 10<sup>th</sup>, 2020
Version 5.1 (Belgium), March 10<sup>th</sup>, 2020
Version 5.0, October 28<sup>th</sup>, 2019
Version 4.0, September 13<sup>th</sup>, 2018
Version 3.0, April 11<sup>th</sup>, 2018

The information contained in this document is the property of Rafael Pharmaceuticals and may not be reproduced, published or disclosed to others without written authorization from Rafael Pharmaceuticals.

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML) Protocol AML003

| Version 8.00 | October 19, 202 |
|--------------|-----------------|
|--------------|-----------------|

### **Table of Content** SPONSOR SIGNATORIES .......ii INVESTIGATOR'S AGREEMENT.......iii Amendment 1 (Version 4.0) ......iv Amendment 2 (Version 5.0) xi Amendment 2.1 (Version 5.1) Amendment 3 (version 6.0) Amendment 4 (version 7.0) 1. PROTOCOL SUMMARY AND SCHEMATIC OF STUDY DESIGN .......34 2. INTRODUCTION: BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE ......44 2.1.1. 2.1.2. 2.1.3. 2.1.4. 2.1.5. 4.2.1. 4.2.2. 4.2.3. Exploratory Endpoints 80 5. STUDY PARTICIPATION AND WITHDRAWAL......81 Exclusion Criteria 83 5.3.1. Definition of Females of Childbearing Potential 86 5.3.2. Acceptable Methods of Effective Contraception .......87 5.3.3. Contraception Methods for Male Patients 87 5.3.4. Unacceptable Methods of Birth Control for Male and Female Patients .......87

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML) Protocol AML003

| Version 8.00 | | October 19, 2020 |
|---|---|---|
| 5.5. Par | ticipant Discontinuation from Treatment or Termination from Study | |
| 5.5.1. | | |
| 5.5.2. | Criteria for Replacing Patients | 90 |
| 5.6. Pre | emature Termination or Suspension of Study | 90 |
| 6. STUD | Y AGENT | 91 |
| 6.1. Stu | dy Agent and Control Description, Formulation, Appearance, Packaging, and | Labeling91 |
| 6.1.1. | High Dose Cytarabine and Mitoxantrone: | 91 |
| 6.1.2. | Mitoxantrone, Etoposide and Cytarabine: | 91 |
| 6.1.3. | Fludarabine, Cytarabine and Filgrastim: | 92 |
| 6.2. Pro | oduct Storage and Stability | 92 |
| 6.2.1. | CPI-613® (devimistat) | 92 |
| 6.2.2. | Cytarabine | 92 |
| 6.2.3. | Mitoxantrone | 92 |
| 6.2.4 | Etoposide | 92 |
| 6.2.5 | Fludarabine | 92 |
| 6.2.6. | Filgrastim | 92 |
| 6.3. Pre | paration | 93 |
| 6.3.1. | CPI-613® (devimistat) | 93 |
| 6.3.2. | Cytarabine, Mitoxantrone, Etoposide, Fludarabine and Filgrastim | 94 |
| Should b | e prepared for administration as outlined in the manufacturers' instructions in | locally approved |
| prescribi | ng information | 94 |
| 6.4. Do | sing and Administration | 94 |
| 6.4.1. | CPI-613® (devimistat) | 94 |
| 6.4.2. | Control Group (HAM) and Control Sub-groups (MEC and FLAG) | 95 |
| 6.4.3. | Treatment Arms and Cycles | 96 |
| 6.4.4. | Dose Adjustments/Modifications/Delays | 111 |
| 6.4.5. | Duration of Therapy | 113 |
| 6.5. Stu | dy Agent Accountability Procedures | 113 |
| 7. STUD | Y PROCEDURES AND SCHEDULE | 115 |
| 7.1. Stu | dy Procedures/Evaluations | 115 |
| 7.1.1. | Medical History | 115 |
| 7.1.2. | Medications History | 115 |
| 7.1.3. | Physical Examination | 115 |
| 7.1.4. | Vital Signs | 115 |
| 7.1.5. | ECOG Performance Status | 115 |
| 7.1.6. | Pharmacokinetic Analysis Blood Sampling (CHAM [Arm 1] Only) | 116 |
| 7.1.7. | ECG Analysis | |
| 7.1.8. | Cardiac marker (Troponin I) | |
| 7.1.9. | Administration of Questionnaires / Other Instruments for Patient-Reported O | |
| 7.2. Sta | ndard of Care Study Procedures | |
| | horatory Procedures/Evaluations | |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML) Protocol AML003

|---|---|---|
| 7.3.1. | Clinical Laboratory Evaluations | 126 |
| 7.3.2. | Other Assays | 127 |
| 7.4. Stu | dy Schedule | 128 |
| 7.4.1. | Screening | 128 |
| 7.4.2. | Randomization/Baseline Visit | 130 |
| 7.4.3. | Study Treatment | 131 |
| 7.4.4. | End of Treatment Visit | 131 |
| 7.4.5. | Safety Follow-Up Visit | 131 |
| 7.4.6. | Long-Term Follow-Up Visit | 131 |
| 7.4.7. | End of Study Visit | 132 |
| 7.4.8. | Schedule of Events Tables | 133 |
| 7.5. Cor | ncomitant Medications, Treatments, and Procedures | 168 |
| 7.6. Pro | phylactic Medications, Treatments, and Procedures | 168 |
| 7.7. Res | cue Medications, Treatments, and Procedures | 169 |
| 7.8. Par | ticipant Access to Study Agent at Study Closure | 169 |
| 8. ASSES | SMENT OF SAFETY | 170 |
| 8.1. Spe | cification of Safety Parameters | 170 |
| 8.1.1. | Definition of Adverse Events | 170 |
| 8.1.2. | Definition of Serious Adverse Events | 170 |
| 8.1.3. | Pregnancy | 171 |
| 8.2. Cla | ssification of an Adverse Event | 172 |
| 8.2.1. | Severity of Event | 172 |
| 8.2.2. | Severity of Adverse Events | 172 |
| 8.2.3. | Expectedness | 174 |
| 8.3. Tin | ne Period and Frequency for Event Assessment and Follow-Up | 174 |
| 8.4. Rep | porting Procedures | 175 |
| 8.4.1. | Adverse Event Reporting | 175 |
| 8.4.2. | Serious Adverse Event Reporting | 176 |
| 8.5. Stu | dy Stopping Rules | 177 |
| 8.6. Saf | ety Oversight | 177 |
| 9. STATIS | STICAL CONSIDERATIONS | 178 |
| 9.1. Stat | tistical and Analytical Plans | 178 |
| 9.2. Stat | tistical Hypotheses | 178 |
| 9.3. Ana | alysis Datasets | 178 |
| 9.4. Des | scription of Statistical Methods | 178 |
| 9.4.1. | General Approach | 178 |
| 9.4.2. | Analysis of Primary Efficacy Endpoint | 179 |
| 9.4.3. | Analysis of Secondary Endpoints | 180 |
| 9.4.4. | Handling Missing Data in Efficacy Analyses | 181 |
| 9.4.5. | Safety Analyses | 181 |
| 9.4.6. | Planned Interim Analyses | 181 |
| 9.4.7. | Additional Sub-Group Analyses. | 181 |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML) Protocol AML003

|---|---|
| 9.4.8. Multiple Comparison/Multiplicity | 182 |
| 9.4.9. Other Secondary Objective Analyses | 182 |
| 9.4.10. Exploratory Objective Analyses | 183 |
| 9.5. Blinding Plan for Statistical Analysis | 184 |
| 9.6. Sample Size | 184 |
| 9.7. Measures to Minimize Bias | 185 |
| 9.7.1. Randomization Procedures | 185 |
| 10. QUALITY ASSURANCE AND QUALITY CONTROL | 186 |
| 11. ETHICS/PROTECTION OF HUMAN PATIENTS | 187 |
| 11.1. Ethical Standard | 187 |
| 11.2. Institutional Review Board/Ethics Committee | |
| 11.3. Informed Consent Process | 187 |
| 11.3.1. Consent/Assent and Other Informational Documents Pro | ovided to Patients187 |
| 11.3.2. Consent Procedures and Documentation | 187 |
| 11.4. Participant and Data Confidentiality | 188 |
| 11.5. Research Use of Stored Human Samples, Specimens or Data | 189 |
| 11.6. Future Use of Stored Specimens | |
| 12. DATA HANDLING AND RECORD KEEPING | 190 |
| 12.1. Data Collection and Management Responsibilities | |
| 12.2. Study Records Retention | |
| 12.3. Protocol Deviations | 190 |
| 12.4. Publication and Data Sharing Policy | 191 |
| 13. STUDY ADMINISTRATION | |
| 13.1. Study Leadership | 192 |
| 14. CONFLICT OF INTEREST POLICY | |
| 15. LITERATURE REFERENCES | 194 |
| 16. APPENDIX A | 196 |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


## LIST OF ABBREVIATIONS

| AE | Adverse Events |
|---|---|
| ALP | |
| ALT | Alkaline Phosphatase |
| AML | Alanine Aminotransferase |
| ANC | Acute Myeloid Leukemia Absolute Neutrophil Count |
| AST | Aspartate Aminotransferase |
| ATP | 1 |
| | Adenosine Triphosphate |
| AUC | Area Under the Plasma Concentration-Time Curve |
| AUCinf | Area Under the Plasma Concentration-Time Curve from Time Zero |
| | Extrapolated to Infinite Time |
| AUC <sub>0-t</sub> | Area Under the Plasma Concentration-Time Curve from Time Zero to the Time |
| DM | of the Last Quantifiable Concentration |
| BM | Bone Marrow |
| BP | Blood Pressure |
| BSA | Body Surface Area |
| BUN | Blood Urea Nitrogen |
| CCAAT | Cytosine-cytosine-adenosine-adenosine-thymidine |
| CEBPa | CCAAT Enhancer Binding Protein A |
| CFR | Code of Federal Regulations |
| СНАМ | CPI-613® (devimistat) in Combination with High Dose Cytarabine and |
| | Mitoxantrone |
| CI | Confidence Interval |
| CL | Apparent Total Body Clearance |
| CrCl | Creatinine Clearance |
| Cmax | The Maximum (Peak) Plasma Drug Concentration |
| Cmin | The Minimum (Trough) Plasma Drug Concentration |
| CMH | Cochran-Mantel-Haenszel |
| CNS | Central Nervous System |
| CR | Complete Remission |
| CRh | CR (Complete Remission) with Partial Hematologic Recovery |
| Cri | CR (Complete Remission) with Incomplete Recovery |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTEP | Cancer Therapy Evaluation Program |
| CTnT | Cardiac Troponin T |
| D5W | Dextrose 5% in Water |
| DEHP | Diethylhexyl Phthalate |
| DMC | Data Monitoring Committee |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EF | Ejection Fraction |
| EORTC QLQ | European Organization for Research and Treatment of Cancer Quality of Life Questionnaire |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


| Version 8.00 | October 19, 2020 | ) |
|--------------|----------------------------------------------------|---|
| EOS | End-of-Study | |
| EOT | End-of-Treatment | |
| FDA | Food and Drug Administration | |
| FLAG | Fludarabine, Cytarabine, and Filgrastim | |
| Flt3 | FMS-Like Tyrosine Kinase 3 | |
| FSH | Follicle Stimulating Hormone | |
| GCP | Good Clinical Practice | |
| GLP | Good Laboratory Practice | |
| GMP | Good Manufacturing Practice | |
| HAM | High Dose Cytarabine and Mitoxantrone | |
| HAMA or HM | High Dose Cytarabine + Mitoxantrone + Asparaginase | |
| hERG | The Human Ether-À-Go-Go-Related Gene | |
| HiDAC | High Dose Cytarabine | |
| HM | High Dose Cytarabine + Mitoxantrone + Asparaginase | |
| HR | Heart Rate | |
| HSCT | Hematopoietic Stem Cell Transplantation | |
| 5-HT | 5-Hydroxytryptamine | |
| IB | Investigator's Brochure | |
| IC50 | The Half Maximal Inhibitory Concentration | |
| ICF | Informed Consent Form | |
| ICH | International Council for Harmonization | |
| IDH1/2 | Isocitrate Dehydrogenase 1 and 2 | |
| IHC | Immunohistochemistry | |
| INR | International Normalized Ratio | |
| IRB | Institutional Review Board | |
| ITD | Internal Tandem Duplication | |
| ITT | Intent-To-Treat | |
| IUD | Intrauterine Device | |
| IUS | Intrauterine Hormonal-Releasing System | |
| IV | Intravenous | |
| IWRS | Interactive Web Response Systems | |
| KGDH | Alpha-Ketoglutarate Dehydrogenase | |
| L-T | Long-Term | |
| LVEF | Left Ventricular Ejection Fraction | |
| MAP | Mean Arterial Pressure | |
| MEC | Mitoxantrone, Etoposide and Cytarabine | |
| MedDRA | Medical Dictionary for Regulatory Activities | |
| MID | Minimal (Clinical) Important Difference | |
| MLFS | Morphological Leukemia-Free State | |
| MRI | Magnetic Resonance Imaging | |
| MTD | Maximum Tolerated Dose | |
| MUGA | Multigated Acquisition Scan | |
| NA | North American | |
| NCCN | National Comprehensive Cancer Network | |
| NCI | National Cancer Institute | |
| NOS | Not Otherwise Specified | |
| ORR | Overall Response Rate | |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003

<u>Version 8.00</u> October 19, 2020

|---|---|
| OS | Overall Survival |
| PDH | Pyruvate Dehydrogenase |
| PK | Pharmacokinetic(s) |
| pKa | Dissociation Constant |
| PP | Per Protocol |
| PR | Partial Remission |
| PRO | Patient-Reported Outcome |
| PS | Performance Score |
| PT | Prothrombin Time |
| PTT | Partial Thromboplastin Time |
| Q12h | Twice a Day with 12 hours Interval |
| QC | Quality Control |
| QD | Once a Day |
| QTc | Corrected QT Interval |
| RNA | Ribonucleic Acid |
| ROW | Rest of the World |
| RR | Respiratory Rate |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Stable Disease |
| SFU | Safety Follow-up |
| SGOT | Serum Glutamic Oxaloacetic Transaminase |
| SGPT | Serum Glutamic Pyruvic Transaminase |
| SUSAR | Suspected Unexpected Serious Adverse Reaction(s) |
| T <sub>1/2</sub> | Elimination half-life |
| TEA | Triethanolamine |
| TF | Treatment Failure |
| TKD | Tyrosine kinase domain |
| Time to Reach the Maximum (Peak) Plasma Concentration following D | |
| | Administration |
| TTE | Transthoracic Echocardiogram |
| ULN | Upper Limit of Normal |
| USP | United States Pharmacopeia |
| $V_d$ | Apparent Volume of Distribution |
| WBC | White Blood Cells |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


## 1. PROTOCOL SUMMARY AND SCHEMATIC OF STUDY DESIGN

| Name of Sponsor: | Rafael Pharmaceuticals, Inc. |
|---|---|
| Protocol Number: | AML003 |
| Name and Description of | CPI-613® (devimistat) |
| <b>Investigational Product:</b> | Mechanism of Action: Targets altered metabolism in cancer cells |
| | [Pyruvate Dehydrogenase (PDH) and α-Ketoglutarate |
| | Dehydrogenase (KGDH) Inhibitor] |
| | <b>Dose:</b> 2,000 mg/m <sup>2</sup> /day in Induction and Consolidation Cycles |
| | and 2,500 mg/m <sup>2</sup> /day in Maintenance Cycles |
| | <b>Route of Administration:</b> Intravenous (IV) infusion, 2 hours |
| Title: | Phase III Multicenter Open-Label Randomized Trial to Evaluate |
| | Efficacy and Safety of CPI-613® (devimistat) in Combination |
| | with High Dose Cytarabine and Mitoxantrone (CHAM) |
| | Compared to High Dose Cytarabine and Mitoxantrone (HAM) |
| | therapy and control sub-groups: combination of Mitoxantrone, |
| | Etoposide and Cytarabine (MEC) and combination of |
| | Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older |
| | Patients (≥50 years) with Relapsed/Refractory Acute Myeloid |
| | Leukemia (AML) |
| Study Duration: | Approximately 48 months |
| Participation Duration: | Approximately 12 months |
| Objectives: | Primary Objective: |
| | ■ To determine efficacy of CHAM in terms of complete |
| | remission (CR) and compare with HAM (control). CR will |
| | be determined as per standard response criteria for AML |
| | (Döhner et al. 2017; 129[4]:424-447). |
| | Secondary Objectives: |
| | ■ To determine efficacy of CHAM in terms of overall |
| | survival (OS) and complete remission + complete |
| | remission with partial hematologic recovery (CR+CRh) |
| | as the two key secondary objectives to compare with HAM |
| | (control). The OS and CR+CRh will be determined as per |
| | standard response criteria for AML (Döhner et al. 2017; |
| | 129[4]:424-447). |
| | <ul> <li>Safety: The assessment of safety will be based mainly on</li> </ul> |
| | the frequency of adverse events (AEs) based on the |
| | Common Terminology Criteria for AEs (version 5.0 or |
| | later) grade. Adverse events will be coded according to the |
| | Medical Dictionary for Regulatory Activities (MeDRA |
| | (version 22.0 or higher). The safety outcomes will include |
| | the occurrence of at least one serious AE, of at least one |
| | Grade 3/4 AE, and of at least one AE requiring the |
| | discontinuation of study treatment. Electrocardiogram |
| | QTc intervals and cardiac markers will also be evaluated. |
| | Other Secondary Objectives: |
| | ■ Pharmacokinetics (PK): to evaluate C <sub>max</sub> , C <sub>min</sub> , AUC, |
| | T <sub>1/2</sub> , T <sub>max</sub> , CL and V <sub>d</sub> for both CPI-613 <sup>®</sup> (devimistat) and |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


its metabolites CPI-2850 and CPI-1810. To evaluate Patient-Reported Outcome (PRO) among patients receiving CHAM compared to HAM as per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30).

■ Cancer-associated mutations and/or genetic alterations in bone marrow aspirates/biopsies and/or peripheral blood. Up to 10 unstained slides from baseline and time of disease progression will be collected. These slides will be used for immuno histochemistry staining for PDKs, PDH, KGDH, SOD2 and CD79a. and as a source of material for RNA and whole exome sequencing should the bone marrow aspirate/biopsy material be inadequate.

### **Exploratory Objectives:**

- Gene expression analysis by RNA sequencing for baseline bone marrow aspirate/biopsy samples to validate previously described response signature from the Phase I study (study CCCWFU 22112). Efficacy and safety analyses per gene mutations will also be assessed (may include FLT3, IDH1/2, TP53, CEBPα, NPM1, etc).
- PK/PD analyses for dose/exposure-response on efficacy and safety.
- Patient Survival: 30-day and 60-day mortality after first dose of study-related treatment.

#### **Endpoints:**

### **Primary Endpoint:**

CR

#### **Secondary Endpoints:**

- OS (key secondary)
- CR+CRh (key secondary)
- Safety
- PK
- PRO by EORTC QLQ-C30
- Cancer-associated mutations and/or genetic alterations in bone marrow aspirate/biopsy and/or peripheral blood

# **Exploratory Endpoints:**

- The determination of the positive and negative predictive value of the gene expression signature found from studying patients on study CCCWFU 22112. Efficacy and safety analyses per gene mutations.
- PK/PD analysis for dose/exposure-response will be explored for clinical efficacy and safety.
- Patient Survival: 30-day and 60-day mortality after first dose of study-related treatment.
- Collection of buccal swabs at Screening/Baseline as a source of germline DNA for comparison with DNA obtained from bone marrow aspirate/biopsy samples.

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


#### **Study Design:**

Phase: III

Study Design: open label, multicenter, randomized trial

**Sample Size:** approximately 500

**Study Groups:** 

- **Arm 1:** CPI-613® (devimistat) + High Dose Cytarabine and Mitoxantrone (CHAM)
- Arm 2: Control group 1: High Dose Cytarabine and Mitoxantrone (HAM)
  - Control sub-group 1: Mitoxantrone, Etoposide and Cytarabine (MEC)
  - o **Control sub-group 2:** Fludarabine, Cytarabine, and Filgrastim (FLAG)

Dosing Schedule of Interventions for CHAM arm (Arm 1): Induction Therapy (up to 2 cycles, each cycle: 14 days): Induction Cycle 1 (14-day cycle):

CPI-613<sup>®</sup> (devimistat) (2,000 mg/m<sup>2</sup> over 2 hours as a central line IV infusion): 5 doses, once a day (QD) Days 1 to 5.

## Followed by:

High Dose Cytarabine following completion of CPI-613® (devimistat) infusion (1 g/m² over 3 hours as a central line IV infusion): 5 doses, every 12 hours (Q12h) starting on Day 3 through Day 5. Time between completion of CPI-613® (devimistat) infusion and the start of Cytarabine infusion should be not more than 2 hours.

# Followed by:

■ <u>Mitoxantrone following completion of High dose Cytarabine infusion</u> (6 mg/m² over 15 minutes as a central line IV infusion): 3 doses, QD following the 1<sup>st</sup>, 3<sup>rd</sup> and 5<sup>th</sup> doses of Cytarabine starting on Day 3 through Day 5 (3 doses). Mitoxantrone given as soon as possible, but no later than 2 hours, after completion of each Cytarabine administration.

**Induction Cycle 2** (14-day cycle; based on Day 14 bone marrow aspirate/biopsy results):

- Patients are only eligible to receive full Induction Cycle 2 therapy if they are hemodynamically stable i.e. mean arterial pressure (MAP) > 60 mm Hg (not on pressors or fluid boluses), have maintained an ejection fraction (EF) sufficient to allow treatment with Mitoxantrone and are able to tolerate it in the opinion of the treating Investigator.
- If no nadir marrow is obtained or after full Induction Cycle 2 therapy, a recovery marrow will be obtained when peripheral blood counts are consistent with remission (absolute neutrophil count [ANC] > 1,000/μL, platelets > 100,000/μL and freedom from blood transfusions) or on

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


Day 42 from the most recent chemotherapy, whichever comes first.

If no Day 14 bone marrow aspirate/biopsy is obtained, no Induction Cycle 2 (Full or Abbreviated) will be given.

Note: Sites that do not perform day 14 bone marrow will not perform induction cycle 2 (full or abbreviated) on any patients at that site. Induction Cycle 2 details:

Same as Cycle 1 or an Abbreviated cycle (14-day cycle) as shown below:

 <u>CPI-613® (devimistat)</u> (2,000 mg/m²): 3 doses, QD Days 1 to 3

Followed by:

 High Dose Cytarabine (1 g/m²) following completion of CPI-613<sup>®</sup> (devimistat) infusion: 3 doses, Q12 h starting on Day 2 through Day 3

Followed by:

 Mitoxantrone (6 mg/m²): 2 doses, QD following the 1<sup>st</sup> and 3<sup>rd</sup> doses of Cytarabine

Cycle 2 is administered as soon as possible, but no later than 5 calendar days, following Day 14 bone marrow aspirate/biopsy results.

**Consolidation Therapy** (for responders to induction):

- Abbreviated course as per Induction Cycles described above (up to 2 consolidation cycles).
- Patients must meet study eligibility criteria for organ function and performance status in order to be eligible for consolidation therapy.

Maintenance Therapy (for responders to induction/consolidation for CHAM arm only):

<u>CPI-613® (devimistat) (2,500 mg/m²)</u>: 5 doses, QD Days 1 to 5 (28-day cycle); continued until disease recurrence, availability of stem cell transplant, the advent of intolerable side effects, or patient withdrawal of consent.

<u>NO</u> administration of High Dose Cytarabine and Mitoxantrone in Maintenance Therapy. Patient may move directly into maintenance therapy if not eligible for re-induction or consolidation therapy.

**Dosing Schedule of Interventions for HAM arm (Control group, arm 2):** HAM group is treated identically with the exception of the omission of CPI-613® (devimistat) and no Maintenance Therapy.

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


## Induction Cycle 1 (14-day cycle):

• <u>High Dose Cytarabine</u> (1 g/m<sup>2</sup> over 3 hours as a central line IV infusion): 5 doses, Q12 hours starting on Day 1 through Day 3.

### Followed by:

Mitoxantrone (6 mg/m² over 15 minutes as a central line IV infusion): 3 doses, QD following the 1<sup>st</sup>, 3<sup>rd</sup> and 5<sup>th</sup> doses of Cytarabine starting on Day 1 through Day 3.

Mitoxantrone given as soon as possible, but no later than 2 hours, after completion of each Cytarabine administration.

**Induction Cycle 2** (14-day cycle; based on Day 14 bone marrow aspirate/biopsy results [as described for CHAM Arm 1 above]).

- Patients are only eligible to receive Induction Cycle 2 therapy if they are hemodynamically stable i.e. MAP > 60 mm Hg (not on pressors or fluid boluses), have maintained an EF sufficient to allow treatment with Mitoxantrone and are able to tolerate it in the opinion of the treating Investigator.
- If no nadir marrow is obtained or after Induction Cycle 2 therapy, a recovery marrow will be obtained when peripheral blood counts are consistent with remission (ANC > 1,000/μL, platelets > 100,000/μL and freedom from blood transfusions) or on Day 42 from the most recent chemotherapy, whichever comes first.
- If no Day 14 bone marrow aspirate/biopsy is obtained, no Induction Cycle 2 (Full or Abbreviated) will be given.

#### Abbreviated Induction Cycle 2:

 High Dose Cytarabine at 1 g/m² administered over 3 hours as a central line IV infusion (as per institutional guidelines or package insert instructions) Q12h starting on Day 1 through Day 2 (total of 3 doses).

#### Followed by:

 <u>Mitoxantrone</u> at 6 mg/m<sup>2</sup> administered over 15 minutes as a central line IV infusion after the 1<sup>st</sup> and 3<sup>rd</sup> doses of Cytarabine (total of 2 doses).

#### **Consolidation Therapy** (for responders to induction):

 Abbreviated course as per Induction Cycles described above (up to 2 consolidation cycles).

**Dosing Schedule of Interventions for MEC (Control sub group, arm 2):** MEC sub-group will be treated as per below defined schedule and there is no Maintenance Therapy.

**Induction Cycle 1 and 2 (2, 14 day-cycles)**: Induction cycle 2 based on Day 14 bone marrow aspirate/biopsy results.

 Etoposide 80mg/m<sup>2</sup> over 60 minutes as a central line IV infusion; 6 doses Day 1 though 6

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003

|---|---|
| | <ul> <li>Cytarabine 1000mg/m² over 3 hours as a central line IV infusion: 6 doses, Day 1 through 6</li> <li>Mitoxantrone 6 mg/m² over 30 minutes as a central line IV infusion: 6 dose, Day 1 through 6</li> </ul> |
| | Consolidation Cycle (1 and 2) (for responders to induction): |
| | <ul> <li>Etoposide 80mg/m² over 60 minutes as a central line IV infusion; 6 doses Day 1 though 6</li> <li>Cytarabine 1000mg/m² over 3 hours as a central line IV infusion: 6 doses, Day 1 through 6</li> <li>Mitoxantrone 6 mg/m² over 30 minutes as a central line IV infusion: 6 dose, Day 1 through 6</li> </ul> |
| | <ul> <li>Dosing Schedule of Interventions for FLAG (Control subgroup, arm 2): FLAG sub-group will be treated as per below defined schedule and there is no Maintenance Therapy.</li> <li>Induction Cycle 1 and 2 (2, 14-day cycles): Induction cycle 2 based on Day 14 bone marrow aspirate/biopsy results.</li> <li>Fludarabine 30mg/m²/day over 30 minutes as a central line IV infusion; 5 doses Day 1 though 5</li> <li>Cytarabine 2g/m² over 4 hours as a central line IV infusion; after Fludarabine: 5 doses, Day 1 through 5</li> <li>Filgrastim 5μg/kg/day by SQ or as per institutional guidelines starting from Day 1 through Day 5 and can resume 7 days after completion of chemo until ANC ≥ 0.5mcL Note: Sites performing Day 14 bone marrow should not administer Filgrastim until the bone marrow is complete. </li> </ul> |
| | <ul> <li>Consolidation Cycle 1 and 2 (2 cycles): <ul> <li>Fludarabine 30mg/m²/day over 30 minutes as a central line IV infusion; 5 doses Day 1 though 5</li> <li>Cytarabine 2g/m² over 4 hours as a central line IV infusion: 4 hours after Fludarabine: 5 doses, Day 1 through 5</li> <li>Filgrastim 5μg/kg/day by SQ or as per institutional guidelines starting from Day 1 through Day 5 and can resume 7 days after completion of chemo until ANC ≥ 0.5mcL</li></ul></li></ul> |
| Number of Sites Enrolling participants: | Approximately 90 sites |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

| | Protocol AML003 |
|---|---|
| Population: | <ul> <li>Sample Size: approximately 500</li> </ul> |
| | <ul> <li>Gender: Both male and female</li> </ul> |
| | • Age: $\geq 50$ years |
| | <ul> <li>Demographic Group: All</li> </ul> |
| | <ul> <li>Eastern Cooperative Oncology Board Performance</li> </ul> |
| | Score (ECOG PS): 0-2 |
| | <ul> <li>Geographic Location: United States, Canada, Austria,</li> </ul> |
| | Belgium, Poland, France, Germany, Spain, Italy, |
| | Australia, South Korea, India and potentially other |
| | countries |
| Main Inclusion Criteria: | ■ Males and females age $\geq$ 50 years must have histologically |
| | documented AML that is relapsed from, or refractory to, |
| | prior standard therapies |
| | Refractory is defined as failure to achieve CR or complete |
| | remission with incomplete recovery (CRi) following: |
| | a. At least one cycle of any anthracycline, cytarabine |
| | or fludarabine containing induction regimen or |
| | persistence of disease on a nadir marrow following |
| | at least one cycle of any anthracycline, cytarabine |
| | or fludarabine containing induction regimen |
| | b. Persistent disease after at least 2 cycles of a |
| | • |
| | hypomethylating agent (azacytidine or decitabine) |
| | with or without venetoclax |
| | <ul> <li>Relapse is defined as development of recurrent AML</li> </ul> |
| | (Döhner et al. 2017; 129[4]:424-447) after CR or CRi has |
| | been achieved with a prior chemotherapy or after disease |
| | progression on a hypomethylating agent with or without |
| | venetoclax |
| | <ul> <li>ECOG PS (performance score) 0-2</li> </ul> |
| | ■ Expected survival greater than 3 months |
| Main Exclusion Criteria: | <ul> <li>Patients who have received previous cytotoxic</li> </ul> |
| | chemotherapy treatment for their relapsed or refractory |
| | AML. Treatment with hypomethylating agents (decitabine |
| | or azacytidine) either alone or in combination with |
| | , |
| | Venetoclax are allowed until the day prior to starting of |
| | CHAM or HAM therapy or control sub-groups (MEC and |
| | FLAG). Targeted therapies including FLT3 or IDH1/2 |
| | inhibitors and/or Hydrea and/or venetoclax are allowed. |
| | Targeted therapies and Hydrea may be taken until the day |
| | prior to starting of CHAM or HAM therapy or control sub- |
| | groups (MEC and FLAG). |
| | • Female patients who are pregnant or breastfeeding or |
| | planning to become pregnant or breastfeed during |
| | treatment and for an additional 6 months after the last dose |
| <u> </u> | 1 |

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003

Version 8.00 October 19, 2020 of CHAM or HAM therapy or control sub-groups (MEC and FLAG) (the teratogenic potential of CPI-613® (devimistat) is unknown). Female patients of childbearing potential with a positive pregnancy test assessed by a serum pregnancy test at Screening. Patients receiving any other standard or investigational treatment for AML, or any other investigational agent for any indication within the past 1 week prior to initiation of CPI-613® (devimistat) treatment (the use of Hydrea and/or venetoclax, oral tyrosine kinase inhibitors FLT3 or IDH 1/2 inhibitors are allowed until the day prior to starting CHAM or HAM therapy or control sub-groups (MEC and FLAG). Previous exposure to a hypomethylating agents either alone or in combination with venetoclax is allowed until the day prior to starting of CHAM or HAM therapy or control sub-groups (MEC and FLAG). Patients who have received immunotherapy of any type within the past 1 week prior to initiation of CPI-613® (devimistat) treatment. Requirement for immediate palliative treatment of any kind including minor surgery. Patients who have received a chemotherapy regimen with autologous stem cell support (bone marrow transplantation) within 6 months of starting CHAM or HAM therapy or control sub-groups (MEC and FLAG). Patients who have had allogenic bone marrow transplantation within the last 6 months. Patients who have had an allogenic transplant more than 6 months ago are eligible provided they have no graft vs host disease. **Statistical Methods:** Primary Endpoint – CR The treatment arm will be compared with the control arm in terms of CR. The significance level will be determined using an O'Brien-Fleming type Lan-DeMets boundary for efficacy equal to 0.023, which will be reached if the difference in CR is larger than 8.3%. This requires 500 patients evaluable for response and will take 36 months after randomization. Endpoint for the 1<sup>st</sup> Interim Analysis – CR This will be performed when 125 patients are evaluable for response after randomization. The significance level for efficacy will be 0.0001 and it will be reached if the difference in CR is larger than 26.7%. The significance level for futility is 0.48 and it will be reached if the difference in CR is less than 0.5%.

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613<sup>®</sup> (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003

October 19, 2020 Version 8.00 Endpoint for the 2<sup>nd</sup> Interim Analysis – CR This will be performed when 250 patients are evaluable for response and after randomization. The significance level for efficacy will be 0.006 and it will be reached if the difference in CR is larger than 12.8%. The significance level for futility is 0.21 and it will be reached if the difference in CR is less than 4.9%. Based on each of these interim analyses, if the CR difference is not sufficiently promising, consideration will be given to stopping the trial; otherwise, the trial will proceed. The final analysis will be performed when 500 patients are evaluable for response. This analysis will take place approximately 36 months after the first randomization. The number of events (deaths) required for secondary analysis is 394. For OS, the re-randomization will use a stratified Cox proportional hazard test-statistic. For CR+CRh, the CMH test-statistic will be used. A Data Monitoring Committee will review safety periodically during the study.

Phase III Multicenter Open-Label Randomized Trial to Evaluate Efficacy and Safety of CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone (CHAM) Compared to High Dose Cytarabine and Mitoxantrone (HAM) therapy and control sub-groups: combination of Mitoxantrone, Etoposide and Cytarabine (MEC) and combination of Fludarabine, Cytarabine, and Filgrastim (FLAG) in Older Patients (≥ 50 years) with Relapsed/Refractory Acute Myeloid Leukemia (AML)

Protocol AML003


## Figure 1 Schematic of Study Design



Abbreviations: CHAM: CPI-613® (devimistat) in Combination with High Dose Cytarabine and Mitoxantrone; CR: complete remission; CRh: complete remission with partial hematologic recovery; ECOG PS: Eastern Cooperative Oncology Group Performance Score; EU: European Union; HAM: High Dose Cytarabine and Mitoxantrone; HiDAC: High Dose Cytarabine; HMA: High Dose Cytarabine + Mitoxantrone + Asparaginase; NA: North American; OS: overall survival; ROW; Rest of the World; Mitoxantrone, Etoposide and Cytarabine (MEC); Fludarabine, Cytarabine and Filgrastim (FLAG).